CLINICAL TRIAL: NCT05120011
Title: Effect of Carnitine Supplementation and Resistance Training on Bone Mineral Density
Brief Title: Carnitine Supplementation and Bone Mineral Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Robert Olek, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BW2021/RO
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Carnitine; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carnitine + leucine (Experimental): 1000 mg L-carnitine with 3000 mg L-leucine per day for 24 weeks
  Interventions: Dietary Supplement: L-carnitine; Dietary Supplement: L-leucine
- leucine (Placebo Comparator): 4000 mg L-leucine per day for 24 weeks
  Interventions: Dietary Supplement: L-leucine

INTERVENTIONS:
Dietary Supplement: L-carnitine — L-carnitine-L-tartrate
  Arms: carnitine + leucine
Dietary Supplement: L-leucine — L-leucine

SUMMARY:
The primary aim of the current research project is to explore whether carnitine supplementation and resistance training may prevent decrements in bone mineral density of aged women.

A secondary aim of this project is to investigate the effect of supplementation on body composition and blood markers.

DETAILED DESCRIPTION:
The study includes postmenopausal women. The subjects participate in resistance training (twice a week) for each session consisted of 6 exercises: horizontal seated leg press, seated chest press, leg extension, shoulder press, lat pull-down seated row, seated cable row.

During the 24-weeks training programme participants are supplemented by carnitine with leucine, or leucine alone (placebo).

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal
* lack of restrictions to perform resistance exercises

Exclusion Criteria:

* cardiovascular disease
* liver disease
* kidney disease
* neuromuscular disease
* gastrointestinal disorders (including stomach ulcers and erosions)
* diabetes
* other severe chronic diseases

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density measured by dual-energy X-ray absorptiometry (DXA) | 24 weeks
  Bone mineral density (BMD) of the femoral neck, lumbar vertebrae L1-L4, and total hip determined by Lunar Prodigy Advance DXA (GE, Healthcare, Madison, Wisconsin, USA).

SECONDARY OUTCOMES:
Body Composition: Body Fat Mass, Fat Free Mass, and Skeletal Muscle Mass using a bioelectrical impedance analyzer (InBody720). | 24 weeks
  The InBody720 measures impedance of five segments of the body (each arm, each leg, trunk) at frequencies of 1, 5, 50, 250, 500, and 1000 kHz through the 8-polar tactile-electrode. Based on the impedance, body fat mass, fat free mass, and skeletal muscle mass are calculated.
The circulating markers modification | 24 weeks
  Determination of serum interleukin-6, tumor necrosis factor alpha, C-reactive protein, and plasma trimethylamine N-oxide.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olek, PhD, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Akademia Wychowania Fizycznego, Poznan, Poland

REFERENCES:
- [Derived] Olek RA, Samborowska E, Wisniewski P, Wojtkiewicz P, Wochna K, Zielinski J. Effect of a 3-month L-carnitine supplementation and resistance training program on circulating markers and bone mineral density in postmenopausal women: a randomized controlled trial. Nutr Metab (Lond). 2023 Aug 2;20(1):32. doi: 10.1186/s12986-023-00752-1. PMID 37533033